CLINICAL TRIAL: NCT05945030
Title: Association of Xanthelasma With Sub Clinical Atherosclerosis and Hepatic Fat: A Case Control Prospective Study
Brief Title: Correlation of Xanthelasma With Atherosclerosis, Hepatic Fat and Fibrosis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Diabetes Foundation, India (Other)
Collaborators: National Diabetes Obesity and Cholesterol Foundation (Other)
Responsible Party: Principal Investigator, Dr Anoop Misra, Director, Diabetes Foundation, India
Other Study IDs: 2023-24/01
Record Dates: First submitted 2023-07-03; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Type2diabetes
MeSH Terms: interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- With Xanthelasma: T2DM with Xanthelasma
  Interventions: Other: Clinical Examination
- Without Xanthelasma: T2DM without Xanthelasma

INTERVENTIONS:
Other: Clinical Examination — T2DM patient visiting Fortis CDOC will undergo clinical examination to determine the grade of Xanthelasma.
  Groups: With Xanthelasma

SUMMARY:
Patients with diabetes with clinical feature of Xanthelasma will show increased Atherosclerosis.

Objectives:

Primary

1. To correlate xanthelasma and its severity to pulse wave velocity and atherosclerosis as see in carotid doppler.

   Secondary
2. To correlate xanthelasma to liver fat and fibrosis.

Methodology:

T2DM patient will be recruited from endocrine OPD

1. Clinical History and Examination:

   a. General Physical Examination: Height, weight, waist circumference, hip circumference, BMI, Blood Pressure, Hand grip. Xanthelasma.
2. Biochemical Test: The biochemical analysis will be done using ELISA kit or commercially available kits

   1. Fasting blood Glucose
   2. Haemoglobin A1C: The estimation of average blood sugar level over a period of two to three months will be analysed with the patient's blood sample for haemoglobin A1C based on turbidimetric inhibition immunoassay method (using COBAS 6000 analyser)
   3. Lipid Profile: Fasting samples shall be analysed for lipid profile. Levels of total cholesterol (TC), serum triglyceride (TG) and high-density lipoprotein cholesterol (HDL-c) will be estimated using commercial kits (Randox Laboratory, USA). Value of low-density lipoprotein cholesterol (LDL-c) will be calculated according to Friedewald's equation.
   4. Liver Function Tests: Fasting samples shall be analysed for liver function test. Levels of alkaline phosphate, Aspartate aminotransferase, Alanine aminotransferase and Gamma-glutamyl transferase will be estimated by using commercial kits (based on kinetic method).
3. Assessment of sub-clinical atherosclerosis: Pulse wave velocity and carotid Doppler will be done

   1. Pulse wave velocity: Arterial stiffness indices will be analyzed by measuring carotid femoral pulse wave velocity.
   2. Carotid Doppler: (based on kinetic method)
   3. FibroScan Estimation: It is a medical diagnostic tool. Liver stiffness (LSM in kPa) and controlled attenuation parameter (CAP in dB/m) measurements will be done by transient elastography (FibroScan® 430 Touch, Echosens, FR) in order to quantify severity of liver fibrosis (LSM 7-10 kPa for F1, 10.1-13 for F2 and >13kPa for F≥3

DETAILED DESCRIPTION:
T2DM is a major public health problem in Asian Indians. Asian Indians develop T2DM at a younger age, and progresses faster than in other ethnic groups. As a result, many diabetes complications are more prevalent and in more advanced stages in Asian countries than in other regions. Asian Indians have one of the highest incidence rates of pre-diabetes and T2DM among all major ethnic groups, and the conversion from pre-diabetes to T2DM occurs more rapidly in this population. According to the Indian Council of Medical Research- India diabetes study (57 117 individuals), the prevalence of prediabetes in all 15 states was 7·3%.

Xanthelasma palpebrarum (XP) are yellow plaques that occur most commonly near the inner canthus of the eyelid and are often associated with atherosclerosis, dyslipidaemia, and coronary artery disease. About 50% of patients who develop xanthelasma have lipid disorder. It is commonly seen in patients with: Type II hyperlipidaemia that includes type IIa, also known as familial hypercholesterolemia, and type IIb, which is commonly referred to as familial combined hyperlipidaemia Type IV hyperlipidaemia, which is also known as familial hypertriglyceridemia: - Diabetes mellitus; Hypothyroidism; Those with low levels of HDL; Fatty diet; Excess alcohol intake; Weight gain.

A significant number of cases of xanthelasma palpebrarum are combined with smoking, central obesity, hypertension, diabetes mellitus, and dyslipidemia which are the major risk factors for CAD. Efforts should be made to rule out the same in high-risk xanthelasma subjects.

Patients with type 2 diabetes mellitus (T2DM) have a high cardiovascular risk even at young age. There is a need to assess this increased risk and identify atherosclerosis early so that appropriate measures for risk reduction can be taken. The Investigators aimed to study carotid-femoral pulse wave velocity (Cf-PWV), a non-invasive indicator of atherosclerosis, in patients with diabetes below 50 years of age and its correlation with markers of obesity and other cardiovascular risk factors.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with T2DM
2. Age 25 to 60 years
3. BMI >25 kg/m² to >40 kg/m²
4. Gender- Both (Male & Female)
5. Mild, moderate and severe Xanthelasma (Photograph)

Exclusion Criteria:

1. Alcoholic abuse or other causes of liver dysfunction.
2. Severe end organ damage or chronic diseases: renal/hepatic failure, any malignancy, major systemic illness etc.

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patient with T2DM visiting Fortis CDOC Hospital will be enrolled in 2 groups cases and controls.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-07-30 (Estimated); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
To determine correlation of Xanthelasma with Pulse wave velocity, Carotid Doppler scores and Fibrosis | 12 month
  Patient with T2DM and Xanthelasma have a high risk of atherosclerosis.

CONTACTS AND LOCATIONS:
Overall Officials: Anoop Misra, MD, Principal Investigator — Fortis CDOC Hospital
Locations (1):
- Fortis CDOC Hospital, Delhi, India

IPD SHARING:
Plan to Share IPD: No